CLINICAL TRIAL: NCT06076343
Title: An Integrated Approach to Treatment of People With Borderline Personality Disorder and Their Caregivers
Brief Title: Integrated Intervention for Borderline Personality Disorder and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Roberta Rossi, Principal investigator, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Integrated interventions
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; caregivers; dialectical behavior therapy; biomarkers; emotion dysregulation
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: consecutive recruitment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dialectical behavior therapy/Family Connections (Experimental): Outpatients with a diagnosis of BPD will be assigned to DBT skills-training intervention (6-10 participants per group). Each DBT skills-training group will receive 24 sessions. Family members of people with BPD will be assigned to psychoeducational intervention. Each FC group (10-12 participants) will receive 12 sessions. Each session for BPD patients and for caregivers lasts 1.5 hours and it is conducted by a leader and a co-leader (two trained psychotherapists).
  Interventions: Behavioral: DBT skills-training and Family Connections interventions

INTERVENTIONS:
Behavioral: DBT skills-training and Family Connections interventions — DBT skills-training program includes four modules: 1. Mindufulness, 2. Distress Tolerance, 3. Emotion Regulation, 4. Interpersonal effectiveness.
  FC program includes six modules: 1. Introduction, 2. Family Education, 3. Relationship Mindfulness Skills, 4. Family Environment Skills, 5. Validation Skills, 6. Problem Management Skills.

SUMMARY:
This is a prospective, single-arm, open-label study to assess the impact of a group intervention for patients with borderline personality disorder (BPD) and a psycho-educational intervention for their caregivers. Once participants complete a comprehensive clinical assessment, the study involves the participation of those with a BPD diagnosis in Dialectical Behavior Therapy (DBT) skills training group, integrated with ongoing routine treatments. A battery of questionnaires is administered before and after the DBT skills training to assess emotion dysregulation, BPD symptoms severity and other clinical variables. Simultaneously, caregivers of individuals with BPD take part in the Family Connections (FC) program. This sub-study follows a previous pilot study conducted at the same centre. Family members complete assessment questionnaires at three different time points (i.e., at baseline, at immediately post-intervention and at a 4-month follow-up) in order to evaluate putative positive pre-post changes on burden, grief and other clinical variables. In order to explore biomarkers of BPD and stress-related neurobiological mechanisms, blood samples are collected from the BPD patient group at pre and post intervention. At baseline, a blood sample is also collected to identify stress-related biomarkers among family members.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) has a severe impact on the lives of individuals with this disorder. Also caregivers of individuals with BPD and related conditions often experience higher levels of somatic and psychological distress. Dialectical Behavior Therapy (DBT) has been proven to be an effective treatment for BPD and it has been well documented that also the module of skills training is effective in the reduction of symptoms. Moreover, one of the most well-established programs to support family members of patients with BPD is Family Connections (FC). FC showed beneficial effects on severity of depression, well-being and family functioning. The aim of the present study is threefold: 1. To evaluate the implementation of a DBT skills training program as a complementary intervention in routine health care. 2. To assess pre-post changes resulting from a FC intervention in family members of individuals with BPD and to identify predictors of positive outcomes. 3. To explore potential biomarkers associated with BPD and stress-related neurobiological mechanisms among both BPD patients and their family members. Participants are recruited at the IRCCS Centro San Giovanni di Dio Fatebenefratelli in Brescia. For the DBT skills training, the primary outcome is the reduction of emotion dysregulation. Secondary outcomes encompass measures of depression, anxiety, alexithymia, global psychological distress, global functioning, impulsiveness, interpersonal problems and severity of BPD symptoms. In addition, socio-demographics, trauma history and the presence of non-suicidal self injury or suicide attempts are assessed. Within the FC group, primary endpoints are burden and grief scores, while secondary endpoints include measurements of depression, alexithymia, global psychological distress, family functioning, and feelings of anger. DBT skills training consists of 24 weekly sessions that incorporate two acceptance-oriented skills (mindfulness and distress tolerance) and two change-oriented skills (emotion regulation and interpersonal effectiveness). The FC program, on the other hand, is a 12-week manualized educational and skills-building support program rooted in the principles of DBT, administered in a group setting to family members of individuals with BPD. Group facilitators possess a medical or psychological professional background and have received training in both the DBT and FC programs. In addition to psychological assessments, the study involves the collection of blood samples from the BPD patient group (before and after the intervention). These samples are collected in order to identify potential biomarkers associated with BPD and treatment response, including levels of Brain-Derived Neurotrophic Factor (BDNF), expression of pro-inflammatory cytokines and anti-inflammatory cytokines, and C-reactive Protein levels. Furthermore, the study analyzes stress-related biomarkers such as cortisol levels and investigate epigenetic mechanisms through DNA and miRNA metilations analysis. In the FC group, a baseline blood sample is also collected to explore stress-related biomarkers.

ELIGIBILITY:
DBT intervention:

Inclusion Criteria:

* to be outpatient with a DBP diagnosis according to DSM5
* age between 18 and 50
* written informed consent

Exclusion Criteria:

* bipolar disorder, psychotic disorders, organic mental disorders, mental retardation, current substance dependence

FC intervention:

* being 18 years of age or older
* serving as a caregiver or significant other of an individual diagnosed with BPD providing written consent

Exclusion Criteria:

- to have a self-reported acute mental health condition interfering with group participation at that time

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) (DBT group) | Baseline, immediately post-intervention
  Change in emotion dysregulation scores on the DERS scale (36 items). Total score of the DERS ranges from 36 to 180 with higher scores indicating higher difficulties in emotion dysregulation.
Burden Assessment Scale (BAS) (FC group) | Baseline, immediately post-intervention, 4-month follow-up
  Change in perceived burden of providing ongoing care to individuals with mental health problems scores. Total score of the BAS ranges from 20 to 80, with higher values indicating stronger burden.
Grief Scale (GS) (FC group) | Baseline, immediately post-intervention, 4-month follow-up
  Change in grief associated with having a loved one with mental illness scores. Total score of the GS ranges from 15 to 75 with higher scores indicating more intense experience of grief.

SECONDARY OUTCOMES:
Beck Depression Inventory II (BDI-II) (FC group and DBT group) | Baseline, immediately post-intervention, 4-month follow-up (FC group). Baseline, immediately post-intervention (DBT group)
  Change in depressive symptoms scores. The BDI-II is evaluated on a severity scale ranging from 0-3, with a total score ranging from 0-63 (higher scores reflecting higher levels of depression).
Symptom Check List-90 (SCL-90) (FC group and DBT group) | Baseline, immediately post-intervention, 4-month follow-up (FC group). Baseline, immediately post-intervention (DBT group)
  Change in the global severity index score of the SCL-90 questionnaire. SCL-90 total scores range from 90-360 with higher scores indicating higher psychological problems.
Toronto Alexithymia Scale 20 (TAS-20) (FC group and DBT group) | Baseline, immediately post-intervention, 4-month follow-up (FC group). Baseline, immediately post-intervention (DBT group)
  Change in alexithymia scores. TAS-20 scoring range: 20-100 (higher scores indicating greater impairment in identifying and describing emotions).
State Trait Anger Expression Inventory (STAXI-2) (FC group and DBT group) | Baseline, immediately post-intervention, 4-month follow-up (FC group). Baseline, immediately post-intervention (DBT group)
  Change in anger severity scores as measured with two subscales of the State Trait Anger Expression Inventory (STAXI-2): 1. the Anger Expression-Out (STAXI-2 ER/OUT) sub-scale measures the frequency in the expression of feelings of anger verbally or physically (range 8-32); 2. the Anger Expression-In (STAXI-2 ER/IN) measures how often the participant experiences anger and suppresses it or withholds it instead of expressing it (range 8-32).
Family Functioning Questionnaire (FFQ) (FC group) | Baseline, immediately post-intervention, 4-month follow-up
  Change in family functioning scores. The FFQ is a 24-item questionnaire with higher scores indicating greater occurrence of positive family related behaviors (total score ranges from 24 to 96).
Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) (DBT group) | Baseline, immediately post-intervention
  Change in frequency of adaptive and maladaptive skills. DBT-WCCL is a 59-item self-report measure of skills used in response to difficult situations over the past month. Two subscales are included: DBT skills use and dysfunctional coping that are rated on a scale of 0-3. Higher score indicates more frequent use of adaptive coping strategies.
Zanarini Rating scale for BPD (DBT group) | Baseline, immediately post-intervention
  Change in overall BPD symptoms severity scores. Zanarini Rating scale for BPD total score ranges from 0 to 36, with higher scores indicating greater severity.
Childhood Trauma Questionnaire short form (CTQ-SF) (DBT group) | Baseline
  Assessment of child maltreatment experiences scores. CTQ is a questionnaire consisting of 28 items, of which 25 measure childhood maltreatment. Total scores for the CTQ-SF range from 25 to 125 with higher scores indicating higher maltreatment severity.
Barratt Impulsiveness Scale-11 (BIS-11) (DBT group) | Baseline, immediately post-intervention
  Change in impulsiveness scores. BIS-11 is a 30-item self-report measure of impulsiveness. Total score ranges from 30 to 120. Higher scores reflecting higher levels of impulsiveness.
Inventory of Interpersonal Problems (IIP-47) (DBT group) | Baseline, immediately post-intervention
  Change in interpersonal functioning scores. The IIP-PD-47 questionnaire is a self-report measure comprised of 47 items on a 5-point Likert scale (higher score reflecting higher interpersonal difficulties).
Attachment Style Questionnaire (ASQ) (DBT group) | Baseline
  Assessment of adult attachment styles. ASQ is a 40-item self-report measure assessing five attachment dimensions, and is answered on a 6-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Rossi, psychologist, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy
Locations (1):
- IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, BS, Italy

REFERENCES:
- [Background] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Background] McMain SF, Links PS, Gnam WH, Guimond T, Cardish RJ, Korman L, Streiner DL. A randomized trial of dialectical behavior therapy versus general psychiatric management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1365-74. doi: 10.1176/appi.ajp.2009.09010039. Epub 2009 Sep 15. PMID 19755574
- [Background] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Background] Liljedahl SI, Kleindienst N, Wangby-Lundh M, Lundh LG, Daukantaite D, Fruzzetti AE, Westling S. Family Connections in different settings and intensities for underserved and geographically isolated families: a non-randomised comparison study. Borderline Personal Disord Emot Dysregul. 2019 Aug 26;6:14. doi: 10.1186/s40479-019-0111-6. eCollection 2019. PMID 31463066
- [Background] Linehan MM, Korslund KE, Harned MS, Gallop RJ, Lungu A, Neacsiu AD, McDavid J, Comtois KA, Murray-Gregory AM. Dialectical behavior therapy for high suicide risk in individuals with borderline personality disorder: a randomized clinical trial and component analysis. JAMA Psychiatry. 2015 May;72(5):475-82. doi: 10.1001/jamapsychiatry.2014.3039. PMID 25806661
- [Derived] Lanfredi M, Meloni S, Ferrari C, Fruzzetti AE, Geviti A, Macis A, Vanni G, Perna G, Diaferia G, Pinti M, Occhialini G, Ridolfi ME, Rossi R. Family Connections: The Impact of an Education Program for Carers of Individuals With Borderline Personality Disorder in Italian Mental Health Services. Fam Process. 2025 Mar;64(1):e13098. doi: 10.1111/famp.13098. PMID 39873150